CLINICAL TRIAL: NCT01171313
Title: A Phase 2 Efficacy, Safety and Pharmacokinetic Study of XP21279 BL2 and Sinemet® in Parkinson's Disease Subjects With Motor Fluctuations
Brief Title: A Efficacy, Safety and Pharmacokinetic Study of XP21279 and Sinemet® in Parkinson's Disease Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP-C-069; XenoPort (Other: XenoPort)
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment sequence 1 (Experimental): Subjects will receive XP21279 and carbidopa, Sinemet, placebo for XP21279 and carbidopa, placebo for Sinemet in a randomized sequence.
  Interventions: Drug: XP21279 and carbidopa (experimental); Drug: Sinemet (comparator); Drug: Placebo for XP21279 and carbidopa; Drug: Placebo for Sinemet
- Treatment sequence 2 (Experimental): Subjects will receive XP21279 and carbidopa, Sinemet, placebo for XP21279 and carbidopa, placebo for Sinemet in a randomized sequence.
  Interventions: Drug: XP21279 and carbidopa (experimental); Drug: Sinemet (comparator); Drug: Placebo for XP21279 and carbidopa; Drug: Placebo for Sinemet
- Treatment sequence 3 (Experimental): Subjects will receive XP21279 and carbidopa, Sinemet, placebo for XP21279 and carbidopa, placebo for Sinemet in a randomized sequence.
  Interventions: Drug: XP21279 and carbidopa (experimental); Drug: Sinemet (comparator); Drug: Placebo for XP21279 and carbidopa; Drug: Placebo for Sinemet
- Treatment sequence 4 (Experimental): Subjects will receive XP21279 and carbidopa, Sinemet, placebo for XP21279 and carbidopa, placebo for Sinemet in a randomized sequence.
  Interventions: Drug: XP21279 and carbidopa (experimental); Drug: Sinemet (comparator); Drug: Placebo for XP21279 and carbidopa; Drug: Placebo for Sinemet

INTERVENTIONS:
Drug: XP21279 and carbidopa (experimental) — Eligible subjects entering the study will be randomized into 1 of 4 sequences where they will be dosed XP21279 and Carbidopa
Drug: Sinemet (comparator) — Eligible subjects entering the study will be randomized into 1 of 4 sequences where they will be dosed Sinemet.
Drug: Placebo for XP21279 and carbidopa — Eligible subjects entering the study will be randomized into 1 of 4 sequences where they will be dosed placebo for XP21279 and carbidopa
Drug: Placebo for Sinemet — Eligible subjects entering the study will be randomized into 1 of 4 sequences where they will be dosed placebo for Sinemet

SUMMARY:
The purpose of the study is to assess the efficacy and safety of XP21279/Carbidopa in comparison to Sinemet as well as evaluate the pharmacokinetics (PK) of levodopa after administration of XP21279/Carbidopa and Sinemet and to explore exposure-response relationships in a subset of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have predictable motor fluctuations of the wearing off type, defined by meeting the following criteria based on the on/off diaries recorded over 3 days in the Screening Period:

   * Wearing-off in at least half (50%) of inter-dose intervals between the first and the last daily doses averaged over the 3 diary days, and
   * An average daily "off" time of 2 hours after the first "on" of the day through awake time up to midnight.
2. Subjects must be on one of the following stable QID or 5 times daily regimens for at least 4 weeks prior to Screening: Sinemet® or carbidopa-levodopa, with a total daily dose ranging from 400 mg to 1000 mg of levodopa

Exclusion Criteria:

1. History, signs, or symptoms suggesting the diagnosis of secondary or atypical Parkinsonism.
2. Subject has moderately or severely disabling dyskinesias for greater than 25% of the waking day
3. Subjects who have significant neurological symptoms not accounted for by Parkinson's disease
4. Subjects who are taking Sinemet® CR, Parcopa®, concomitant COMT inhibitors (i.e., entacapone or tolcapone), Stalevo®, or benserazide containing levodopa preparations Madopar® or Prolopa®.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mean daily "off" time at end of double-blind maintenance treatment periods. | 2 weeks

SECONDARY OUTCOMES:
Proportion of responders ("much improved" or "very much improved") on Investigator-rated and patient-rated CGI-I at end of double-blind Maintenance Treatment periods | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan Chen, M.D., Study Director — XenoPort, Inc.
Locations (12):
- United States (12):
  - XenoPort Clinical Site, Phoenix, Arizona
  - XenoPort Clinical Site, Little Rock, Arkansas
  - XenoPort Clinical Site, Long Beach, California
  - XenoPort Clinical Site, Sunnyvale, California
  - XenoPort Clinical Site, Naples, Florida
  - XenoPort Clinical Site, Tampa, Florida
  - XenoPort Clinical Site, Kansas City, Kansas
  - XenoPort Clinical Site, Bingham Farms, Michigan
  - XenoPort Clinical Site, West Bloomfield, Michigan
  - XenoPort Clinical Site, New Brunswick, New Jersey
  - XenoPort Clinical Site, Tulsa, Oklahoma
  - XenoPort Clinical Site, Houston, Texas